CLINICAL TRIAL: NCT05549999
Title: Cultural Adaptation, Validity, and Reliability of the Turkish Version of North Star Ambulatory Assessment
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Güllü AYDIN YAĞCIOĞLU, Research Asisstant, Suleyman Demirel University
Other Study IDs: NSAA-123
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Duchenne Muscular Dystrophy; Ambulation Difficulty; Ambulation Disorder, Neurologic
Keywords: Duchenne Muscular Dystrophy; Ambulation; reliability; validity
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Mobility Limitation; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: North Star Ambulatory Assessment — North Star Ambulatory Assessment is an ambulatory assessment developed specifically for Duchenne Muscular Dystrophy.

SUMMARY:
The aim of this study is to translate the "North Star Ambulatory Assessment (NSAA)" scale into Turkish and make its cultural adaptation and to demonstrate the reliability and validity of the Turkish version in patients with ambulatory DMD. For the translation into Turkish, validity and reliability of the NSAA, necessary permission was obtained from the developer of the questionnaire, Prof. Dr. Francesco Muntoni, via e-mail. In the study, first of all, the translation and cultural adaptation process will be completed, and then reliability-validity studies will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with DMD
* Ambulatory
* Being between the ages of 4-18
* Agreeing to participate in the research voluntarily

Exclusion Criteria:

* Insufficient cooperation with the physiotherapist,
* Have had any injury and/or surgery of the lower extremities in the last 6 months,
* Having neurological problems in addition to DMD. -

Ages: 4 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study population include just ambulatory patients with Duchenne Muscular Dystrophy
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
North Star Ambulatory Assessment | 10 minutes
  The North Star Ambulatory Assessment (NSAA) is a functional scale specifically designed for ambulant boys with DMD. The instrument contains clear and detailed instructions, with item scores varying according to a simple three point criteria, which should allow accurate reproduction by different groups. The scale has also the advantage to be quick to perform and to be suitable for application in young children. The NSAA also includes two timed items, run/walk for 10 meters and rise from the floor. While those times do not influence the score, they can be used to monitor changes over time. Although it was developed to assess ambulatory patients, the NSAA has been widely accepted and used to evaluate ambulatory motor performance in children and young adults with DMD, as well as in patients with other neuromuscular diseases.

SECONDARY OUTCOMES:
Motor Function Measure (MFM) | 20-30 minutes
  MFM, which was valid and reliable in Neuromuscular Diseases, was used for gross motor function assessment. The items in MFM, which evaluate functions in 3 different sections (D1, standing position and transfers; D2, axial and proximal motor function; D3, distal motor function) in 32 items in total, are scored between 0-3. 0; cannot initiate any movement and maintain the starting position, 1; partially completes the exercise, 2; performs the exercise slowly and visibly clumsily, with compensations, 3; performs the exercise in the specified standard pattern. High scores indicate higher motor function and the result is expressed as a percentage of the maximum possible score to enable comparison with other scores
6 meter walking test (6MWT) | 6 minutes
  6MWT is an assessment that was developed by Balke in the 1960s and has validity and reliability for DMD patients. The maximum distance that the patient can walk in 6 minutes is recorded as meters.

CONTACTS AND LOCATIONS:
Overall Officials: Güllü Aydın Yağcıoğlu, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Güllü Aydın Yağcıoğlu, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aydin-Yagcioglu G, Bulut N, Ugur F, Yilmaz O, Alemdaroglu-Gurbuz I. Cultural adaptation, validity and reliability of the Turkish version of north star ambulatory assessment. Acta Neurol Belg. 2025 Feb;125(1):127-132. doi: 10.1007/s13760-024-02670-2. Epub 2024 Oct 22. PMID 39436553